CLINICAL TRIAL: NCT06640075
Title: Co-produced Community Action for Improved Access to Cervical Cancer Screening (Act4CC): a Mixed-methods Study in Rural Areas of the Mifi Health District
Brief Title: Community Co-produced Action for Improved Access to Cervical Cancer Screening in Cameroon
Acronym: Act4CC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Patrick Petignat (Other)
Collaborators: University Hospital, Geneva (Other); Bafoussam Regional Hospital, Cameroon (Unknown); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor-Investigator, Prof. Patrick Petignat, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1020/31/01/2024/CE/CRERSH-OU/V; AO_2023-00019 (Other: Commission cantonale d'éthique de la recherche de Genève)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Intervention Model Description: cluster-randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community co-produced action (Experimental): Participatory workshops will be conducted with community members by a multidisciplinary team with the aim to co-develop a strategy for cervical cancer screening adapted to the local setting (including primary HPV screening, triage of HPV-positive patients and treatment of patients triaged positive).
  Interventions: Other: Community co-produced action
- Standard screening strategy (Active Comparator): Recruitment of study participants will be coordinated centrally at district level (from the Bafoussam Regional Hospital) following procedures previously established in a cervical cancer screening program in the health district of Dschang.
  Interventions: Other: Standard screening strategy

INTERVENTIONS:
Other: Community co-produced action — Participatory workshops will be conducted with community members by a multidisciplinary team with the aim to co-develop a strategy for cervical cancer screening adapted to the local setting (including primary HPV screening, triage of HPV-positive patients and treatment of patients triaged positive). This intervention is referred to as 'community co-produced action'. Possible strategies co-developed may include collaboration with community health workers or local associations, awareness campaigns, development of health education materials, integration of primary HPV screening at local integrated health centers, organization of group transportation to the district screening center, etc.
  Using purposive sampling methods, approximately 15 participants will be invited to take part in the workshops in each health area of the intervention, including approximately 3 health care providers, 3 community health workers or members of women's associations, 3 men and 6 eligible women for screening.
  Arms: Community co-produced action
Other: Standard screening strategy — Recruitment of study participants will be coordinated centrally at district level (from the Bafoussam Regional Hospital) following procedures previously established in a cervical cancer screening program in the health district of Dschang. This standard procedure includes the training of 2 community health workers (CHW) by health area to raise awareness around cervical cancer. After an initial theoretical and practical training in cervical cancer prevention, CHWs recruit women by going door-to-door or through community meetings in their respective health areas. Through a system of nominal invitation vouchers distributed to eligible women, CHWs receive a financial incentive for each woman that shows up for cervical cancer screening. Twice a year, CHWs of all health areas are invited to a feedback session to discuss difficulties encountered on the field and propose solutions to face any identified challenges.
  Arms: Standard screening strategy

SUMMARY:
Background - The burden of cervical cancer is unequally distributed globally, with over 90% of deaths occurring in low- and middle-income countries (LMICs), mainly due to insufficient uptake of preventive measures such as screening. In 2020, the World Health Organization launched a global initiative for the worldwide elimination of cervical cancer as a public health issue, setting a target of 70% of women screened with a high-performance test. In Cameroon, this target is far from being reached, and rural communities are disproportionately affected by low uptake of screening services. Recently, a new cervical cancer screening program has launched in the Bafoussam Regional Hospital, in the capital of the Mifi Health District, as part of a larger research project. To develop a context-specific strategy improving access to screening for women living in rural areas of the district, the active participation of community members for the co-development and implementation of local strategies for cervical cancer screening may be key to improving population screening coverage.

Objective - The aim of this study is to evaluate the use of community co-produced action (CCA) for the development and implementation of HPV-based cervical cancer screening strategies compared to a traditional hospital-based approach in rural areas of the Mifi Health District in Cameroon.

Methods - Using a cluster-randomized study design, participatory workshops with community members will be led in 7 rural health areas assigned to the intervention arm, with the aim of codeveloping local strategies for HPV-based cervical cancer screening adapted to the setting. The co-produced strategies may include raising awareness among eligible women (aged 30-49 years, or 25-49 years if HIV-positive), as well as facilitating access to screening tests, results and follow-up. Women living in one of the 7 health areas assigned to the control arm will be invited by community health workers to undergo screening at the Bafoussam Regional Hospital. In both study arms, screened women will be included in the GENOVA study, a cervical cancer screening trial offering free-of- charge HPV testing followed by triage by visual inspection or genotyping for HPV-positive women, and free treatment according to triage results. CCA will be evaluated by assessing its effectiveness for screening uptake. Screening coverage among eligible women will be estimated during one year after implementation of screening strategies in both study arms, based on population statistics provided by the Mifi health district for each health area.

Expected results - Developing context-sensitive solutions to cervical cancer screening through a community-based participatory approach in rural areas of the Mifi health district is expected to improve screening participation rate.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-49 years old (25-49 years old if HIV-positive)
* Residency in one of the 14 rural health areas of Mifi health district
* Ability to give signed informed consent

Exclusion Criteria:

* known cervical cancer
* symptoms compatible with cervical cancer
* previous hysterectomy
* terminal disease other than cervical cancer
* cervical cancer screening test in the last 5 years (3 years if HIV-positive)
* pregnancy at the time of screening
* lack of discernment capacity

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-04-13 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of women having completed screening for cervical cancer | Within 12 months after implementation of the screening strategy at health-area level
  Coverage rate of complete screening (defined as an HPV test +/- triage for HPV-positive women) among the eligible population in both study arms within 12 months.

SECONDARY OUTCOMES:
Number of women having completed primary screening | Within 12 months after implementation of the screening strategy at health-area level
  Rate of primary screening (HPV test) among the eligible population in both study arms.
Number of HPV-positive women having completed triage and treatment when necessary | Within 3 months after primary screening (HPV test)
  Proportion of women with positive primary screening who proceed to completing triage and treatment (when needed) in both study arms
Number of HPV-positive women attending a follow-up visit at 12 months | From 11 to 15 months after primary screening
  Proportion of HPV-positive women who attend the follow-up visit at 12 months after primary screening (HPV test) in both study arms
Number of women with different sociodemographic characteristics | At enrollment
  Distribution of sociodemographic characteristics among screened women in both study arms

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Petignat, PD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Bafoussam Regional Hospital, Bafoussam, Mifi, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will be made available on an open-access repository alongside a data dictionary. All IPD used in the results publication will be published.
Supporting Information: Study Protocol
Time Frame: Upon result publication and for a minimum of 10 years.
Access Criteria: The anonymized IPD will be made available on an open-access data repository.
URL: https://yareta.unige.ch/home